CLINICAL TRIAL: NCT01706380
Title: A Randomized Controlled Trial of Interactive Voice Response With and Without Personal Feedback in the Treatment of Adolescents With Substance Use Disorders
Brief Title: 3M Study - Maria Malmö Mobile Telephone Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Anders C Håkansson, MD, PhD, Region Skane
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3M Study
Record Dates: First submitted 2012-10-08; First posted 2012-10-15 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Substance Use Disorders
Keywords: Substance use disorders; Adolescents; Retention; Mobile telephone; Follow-up; Interactive voice response
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interactive voice response with personal feedback (Experimental): Interactive voice response follows the client twice weekly for 3 months with respect to symptoms and substance use, in both arms. This intervention group also receives a personalized and automated feedback describing whether the symptom status of the patient is better, worse or equal, compared to the preceding follow-up.
  Interventions: Behavioral: Interactive voice response with personal feedback
- Interactive voice response without personal feedback (Active Comparator): This control group is also followed with identical interactive voice response follow-up, addressing symptoms and substance use, but without the personal feedback.
  Interventions: Behavioral: Interactive voice response without personal feedback

INTERVENTIONS:
Behavioral: Interactive voice response with personal feedback — Personal feedback is given at the end of each automated telephone follow-up call, and reports back to the patient whether his och her symptom status is better, worse or equal, compared to the previous telephone call.
  Arms: Interactive voice response with personal feedback
Behavioral: Interactive voice response without personal feedback — Control condition. Identical follow-up but without personal feedback.
  Arms: Interactive voice response without personal feedback

SUMMARY:
The present study, in an out-patient setting for substance use treatment in adolescents, examines the effect on treatment retention of a mobile telephone follow-up technique (interactive voice response), with or without personal feedback. Subjects in treatment for substance use disorders will be followed by automated mobile telephone contact with questions about psychiatric symptoms and substance use, and the investigators hypothesize that this technique, including a personal feedback reporting back to the client whether his or her status is changing in one way or another, may increase the treatment retention, possibly by means of an intensified treatment contact.

ELIGIBILITY:
Inclusion Criteria:

* Patient applying for substance use disorder treatment at out-patient facility Maria Malmö, Malmö, Sweden, who are less than 25 years old and who provide written informed consent to participate in the study.

Exclusion Criteria:

* Patients who do not provide written informed consent to the study, or whose psychiatric condition or language difficulties make it impossible for them to understand patient information and give informed consent to the study.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 73 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Retention in substance use disorder treatment | 3 months
  Duration of retention in treatment and whether the client remains in treatment at 3 months or not.

SECONDARY OUTCOMES:
Improvement in substance use | 3 months
  Do patients in the intervention group improve more than in the control group, with respect to substance use (alcohol/drug use), during the duration of the interactive voice response intervention?
Improvements in psychiatric symptoms | 3 months
  Do patients in the intervention group improve more than in the control group, with respect to psychiatric symptoms, during the duration of the interactive voice response intervention?

OTHER OUTCOMES:
Clinical course with respect to emergency visits | 12 months
Clinical course with respect to hospitalizations | 12 months
Clinical course with respect to repeated treatment episodes | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Malmö, Dept of Psychiatry Skane and City of Malmö, Sweden, Malmo, Skåne County, Sweden